CLINICAL TRIAL: NCT03590340
Title: Randomized, Double-Blind, Placebo-Controlled, Regimen Optimization Study of a Radiation-Attenuated Plasmodium Falciparum (Pf) Sporozoite Vaccine (PfSPZ Vaccine) in Equatoguinean Adults
Brief Title: Regimen Optimization Trial of PfSPZ Vaccine in Equatorial Guinea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanaria Inc. (Industry)
Collaborators: Ifakara Health Institute (Other); Swiss Tropical & Public Health Institute (Other); Government of Equatorial Guinea (Other Government); Noble Oil Services (Industry); Marathon Oil Corporation (Industry); Atlantic Methanol Production Company (Unknown); Equatorial Guinea (EG) liquefied natural gas (LNG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EGSPZV3
Record Dates: First submitted 2018-06-12; First posted 2018-07-18 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; PfSPZ Vaccine; PfSPZ Challenge (NF54); CHMI
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Group 1a (PfSPZ Vaccine) (Experimental): Group 1a: subjects (n=21) will receive four doses of PfSPZ Vaccine (9.0 x 10^5 PfSPZ/dose) on Days 1, 3, 5, and 7 as a prime, followed by a boost of 9.0x10^5 PfSPZ Vaccine on Day 113.
  Controlled human malaria infection (CHMI) with PfSPZ Challenge (NF54) will be administered 8 weeks after the last boost dose by DVI injection.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (for CHMI)
- Group 2a (PfSPZ Vaccine) (Experimental): Group 2a: subjects (n=21) will receive four doses of PfSPZ Vaccine (9.0 x 10^5 PfSPZ/dose) on Days 1, 3, 5, and 7 as a prime.
  CHMI with PfSPZ Challenge (NF54) will be administered 8 weeks after the last prime dose by DVI injection.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (for CHMI)
- Group 3a (PfSPZ Vaccine) (Experimental): Group 3a: subjects (n=21) will receive four doses of PfSPZ Vaccine (9.0 x 10^5 PfSPZ/dose) on Days 1, 3, 5, and 7 as a prime, followed by a boost of 9.0x10^5 PfSPZ Vaccine on Day 29.
  CHMI with PfSPZ Challenge (NF54) will be administered 8 weeks after the last boost dose by DVI injection.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (for CHMI)
- Group 4a (PfSPZ Vaccine) (Experimental): Group 4a: subjects (n=21) will receive two doses of PfSPZ Vaccine (9.0 x 10^5 PfSPZ/dose) on Days 1 and 8 as a prime, followed by a boost of 9.0x10^5 PfSPZ Vaccine on Day 29.
  CHMI with PfSPZ Challenge (NF54) will be administered 8 weeks after the last boost dose by DVI injection.
  Interventions: Biological: PfSPZ Vaccine; Biological: PfSPZ Challenge (for CHMI)
- Group 1b (NS) (Placebo Comparator): Group 1b: subjects (n=5) will receive normal saline (NS) placebo on Days 1, 3, 5, 7, and 113.
  CHMI with PfSPZ Challenge (NF54) will be administered 8 weeks after the last immunization by DVI.
  Interventions: Other: Normal saline; Biological: PfSPZ Challenge (for CHMI)
- Group 2b (NS) (Placebo Comparator): Group 2b: subjects (n=5) will receive NS placebo on Days 1, 3, 5, and 7.
  CHMI with PfSPZ Challenge (NF54) will be administered 8 weeks after the last immunization by DVI.
  Interventions: Other: Normal saline; Biological: PfSPZ Challenge (for CHMI)
- Group 3b (NS) (Placebo Comparator): Group 3b: subjects (n=5) will receive NS placebo on Days 1, 3, 5, 7, and 29.
  CHMI with PfSPZ Challenge (NF54) will be administered 8 weeks after the last immunization by DVI.
  Interventions: Other: Normal saline; Biological: PfSPZ Challenge (for CHMI)
- Group 4b (NS) (Placebo Comparator): Group 4b: subjects (n=5) will receive NS placebo on Days 1 and 8.
  CHMI with PfSPZ Challenge (NF54) will be administered 8 weeks after the last immunization by DVI.
  Interventions: Other: Normal saline; Biological: PfSPZ Challenge (for CHMI)

INTERVENTIONS:
Biological: PfSPZ Vaccine — Metabolically active, non-replicating, radiation attenuated, aseptic, purified, cryopreserved NF54 P. falciparum (Pf) sporozoites (PfSPZ Vaccine)
  Arms: Group 1a (PfSPZ Vaccine); Group 2a (PfSPZ Vaccine); Group 3a (PfSPZ Vaccine); Group 4a (PfSPZ Vaccine)
Other: Normal saline — Normal saline is 0.9% sodium chloride
  Arms: Group 1b (NS); Group 2b (NS); Group 3b (NS); Group 4b (NS)
Biological: PfSPZ Challenge (for CHMI) — Live, infectious, aseptic, purified, vialed, cryopreserved, Plasmodium falciparum sporozoites, strain NF54

SUMMARY:
This is a phase 1, randomized regimen optimization study of PfSPZ Vaccine in healthy Equatoguinean volunteers to determine if a condensed, rapid immunization regimen is safe and efficacious. Four different regimens 4 weeks or less in duration will be evaluated for safety, tolerability, immunogenicity, and protective efficacy in comparison to a gold standard 16-week regimen.

DETAILED DESCRIPTION:
This double-blind, placebo-controlled clinical trial will be conducted in 104 Equatoguinean healthy men and women 18-45 years of age divided into four groups of 26 subjects receiving one of four dosing regimens. The study is designed to test the hypothesis that 2 or 4 doses of 9x10^5 PfSPZ of PfSPZ Vaccine administered by direct venous inoculation (DVI) over 6-7 days as the priming immunization, with or without a boosting immunization at 4 or 16 weeks after the last priming dose, will (1) be safe and well tolerated; and (2) induce immunity leading to protection against homologous controlled human malaria infection (CHMI) performed at 8 weeks after the final immunization by DVI injection of PfSPZ Challenge. The first regimen will test the radiation-attenuated whole sporozoite PfSPZ Vaccine in a dose of 9.0x10^5 administered by DVI with four priming immunizations followed by a boost after 16 weeks. The second regimen will follow the same dosing and administering schedule, but without the boost after 16 weeks to study if a boost may be necessary. The third regimen will follow the first regimen with the interval duration to the boost shortened to only 4 weeks. In the fourth and final regimen, the vaccine will be administered two times instead of four followed by a boost in 4 weeks to evaluate if two priming immunizations will be sufficient to confer protection. In summary:

* Group 1: 21 subjects will receive 9.0x10^5 PfPSZ and 5 subjects will receive normal saline (NS) placebo on Days 1, 3, 5, 7, and 113.
* Group 2: 21 subjects will receive 9.0x10^5 PfPSZ and 5 subjects will receive NS on Days 1, 3, 5, and 7.
* Group 3: 21 subjects will receive 9.0x10^5 PfPSZ and 5 subjects will receive NS on Days 1, 3, 5, 7, and 29.
* Group 4: 21 subjects will receive 9.0x10^5 PfPSZ and 5 subjects will receive NS on Days 1 and 8.

The safety and tolerability of each regimen will be measured by recording (1) solicited and unsolicited adverse events, (2) immunogenicity by assessing humoral and cellular immune responses pre- and post-vaccination, and (3) vaccine efficacy (VE) by measuring protection against homologous CHMI administered by DVI of PfSPZ Challenge (NF54) at 8 weeks post-final vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and non-pregnant/non-lactating females, age 18 to 45 years at time of enrollment.
2. Provision of signed and dated informed consent form.
3. Demonstrate understanding of the study by responding correctly to 10 out of 10 true/false statements about the trial (a maximum of two additional attempts will be granted for those who fail to respond correctly to all true/false statements in their first attempt).
4. Stated availability and willingness to comply with all study procedures and visits for the duration of the trial, including the required vaccination and post-CHMI ward observation period.
5. Able to understand and communicate in Spanish, the national language of Equatorial Guinea
6. Be in good general health as evidenced by medical history, screening physical examination and laboratory findings.
7. Females of child bearing potential must agree to use injectable medroxyprogesterone for at least 4 weeks prior to enrollment and agree to continue to use medroxyprogesterone during the entire study period.
8. Female subjects must not be pregnant (as demonstrated by a negative urine pregnancy test) at enrollment and prior to each immunization.
9. Body Mass Index (BMI) of 18 to 30 kg/m2.
10. At least one year of residence on Bioko Island, Equatorial Guinea, and living close enough to Baney Clinical Research Center and Sampaka Hospital to be able to attend the required appointments at the study center.
11. Agree to release medical information and inform a study doctor about contraindications for participation in the study.
12. Willingness to be attended to by a study doctor and take all medications prescribed during the study period.
13. Agree to provide contact information of a third-party household member or close friend to the study team.
14. Agree not to participate in another clinical trial during the study period.
15. Agree not to donate blood during the study period.
16. Willing to undergo HIV, hepatitis B (HBV) and hepatitis C (HCV) tests.
17. Reachable by telephone for adverse event review.

Exclusion Criteria:

1. Known allergic reactions to components of PfSPZ Vaccine, PfSPZ Challenge, or artemether-lumefantrine (AL).
2. Having received an investigational malaria vaccine in the last 5 years.
3. Having received any non-live vaccine in the 14 days prior to enrollment, any live vaccine in the 28 days prior to enrollment or three or more of any type of vaccine in the four months prior to enrollment.
4. Participation in any other clinical study involving investigational medicinal products including malaria drugs within 30 days prior to enrollment.
5. History of arrhythmias, prolonged QT-interval or other cardiac disease, or clinically significant abnormalities on electrocardiogram (ECG) at screening.
6. History of non-febrile seizures or complex febrile seizures.
7. History of cardiac disease in a 1st or 2nd degree relative when <50 years of age.
8. A chronic illness including diabetes mellitus, cancer, HIV/AIDS, tuberculosis.
9. History of illicit drug or alcohol use that interferes with normal social function.
10. The use of chronic immunosuppressive drugs or other immune modifying drugs within three months of study onset (inhaled and topical corticosteroids are allowed) and during the study period.
11. Any clinically significant deviation from the normal range in biochemistry, hematology or urinalysis tests.
12. Positive HIV, hepatitis B virus or hepatitis C virus serologic tests.
13. Signs and symptoms of tuberculosis (e.g., chronic cough, night sweats, chronic fever, enlarged lymph nodes, unintended weight loss), or risk factors in an otherwise healthy person in combination with a positive tuberculin skin test (TST).
14. Symptoms, physical signs and/or laboratory values suggestive of systemic disorders including renal, hepatic, blood, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteer.
15. Any medical, psychiatric, social or occupational condition or situation that, in the judgment of the PI, impairs the volunteer's ability to give informed consent, increases the risk to the volunteer of participation in the study, affects the ability of the volunteer to participate fully in the study, or might negatively impact the quality, consistency or interpretation of data derived from their participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Incidence and type of Adverse Events (AEs) | Day of first immunization until 1 year
  1. Occurrence of solicited local AEs during priming vaccination and a 3-day surveillance period after priming and boost vaccinations.
  2. Occurrence of solicited systemic AEs during priming vaccination and a 7-day surveillance period after priming and boost vaccinations.
  3. Occurrence of unsolicited AEs during priming vaccination and a 14-day surveillance period after priming and boost vaccinations.
  4. Occurrence of serious adverse events (SAEs) during the study.

SECONDARY OUTCOMES:
Proportion of volunteers who become parasitemic will be recorded, detected by thick blood smear microscopy (TBS) and/ or quantitative real time polymerase chain reaction (qPCR) | Post first immunization uptil 56 days post-CHMI
  1. Development of Pf parasitemia by TBS following CHMI
  2. Development of Pf parasitemia by qPCR following CHM
Level of Antibodies against Pf proteins in volunteer sera | Post first immunization uptil 56 days post-CHMI
  1. Antibody titres to pre-erythrocytic stage and erythrocytic stage antigens[PfCSP, PfLSA-1, PfEBA-175 , PfMSP-1, PfMSP-5, EXP-1] by ELISA
  2. Antibody titres to Pf sporozoites, asexual and sexual erythrocytic stage parasites by IFA.
  3. Analysis of antibodies to proteins in the Pf proteome array chip.
Inhibitory Capacity of Volunteer Sera against in vitro Sporozoite Invasion of Hepatocytes | Post first immunization uptil 56 days post-CHMI
  Capacity of sera from immunized volunteers to inhibit sporozoite invasion (ISI) of hepatocytes in vitro by ISI assay

CONTACTS AND LOCATIONS:
Overall Officials: Said Jongo, MD, MMed, Principal Investigator — Ifakara Health Institute
Locations (1):
- Baney Clinical Research Center, Santiago de Baney, Bioko Island, Equatorial Guinea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mpina M, Stabler TC, Schindler T, Raso J, Deal A, Acuche Pupu L, Nyakarungu E, Del Carmen Ovono Davis M, Urbano V, Mtoro A, Hamad A, Lopez MSA, Pasialo B, Eyang MAO, Rivas MR, Falla CC, Garcia GA, Momo JC, Chuquiyauri R, Saverino E, Preston Church LW, Kim Lee Sim B, Manguire B, Tanner M, Maas C, Abdulla S, Billingsley PF, Hoffman SL, Jongo S, Richie TL, Daubenberger CA. Diagnostic performance and comparison of ultrasensitive and conventional rapid diagnostic test, thick blood smear and quantitative PCR for detection of low-density Plasmodium falciparum infections during a controlled human malaria infection study in Equatorial Guinea. Malar J. 2022 Mar 24;21(1):99. doi: 10.1186/s12936-022-04103-y. PMID 35331251